CLINICAL TRIAL: NCT06455449
Title: A Multicenter, Parallel-group, Double-blind, 2-Arm, Phase III Study to Investigate the Efficacy and Safety of Anifrolumab Administered as Subcutaneous Injection and Added to Standard of Care Compared With Placebo Added to Standard of Care in Adult Participants With Idiopathic Inflammatory Myopathies (Polymyositis and Dermatomyositis)
Brief Title: A Study to Investigate the Efficacy and Safety of Anifrolumab Administered as Subcutaneous Injection and Added to Standard of Care Compared With Placebo Added to Standard of Care in Adult Participants With Idiopathic Inflammatory Myopathies (Polymyositis and Dermatomyositis)
Acronym: JASMINE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3463C00003
Record Dates: First submitted 2023-09-28; First posted 2024-06-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Polymyositis, Dermatomyositis
Keywords: Polymyositis; Dermatomyositis; anifrolumab
MeSH Terms: conditions — Dermatomyositis; Polymyositis | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (subcutaneous weekly injection) (Experimental): Anifrolumab subcutaneous injection once weekly
  Interventions: Combination Product: Anifrolumab (blinded); Combination Product: Anifrolumab (unblinded, open label)
- Placebo (subcutaneous weekly injection) (Placebo Comparator): Matched placebo control subcutaneous injection once weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Anifrolumab (blinded) — Anifrolumab treatment delivered subcutaneously, once weekly for 52 weeks
  Other Names: Treatment arm (blinded)
  Arms: Anifrolumab (subcutaneous weekly injection)
Other: Placebo — Matched placebo delivered subcutaneously, once weekly for 52 weeks
  Other Names: Placebo arm (blinded)
  Arms: Placebo (subcutaneous weekly injection)
Combination Product: Anifrolumab (unblinded, open label) — At Week 52, all study participants on anifrolumab or placebo will receive open label anifrolumab once weekly for an additional 52 weeks
  Other Names: treatment arm (unblinded)
  Arms: Anifrolumab (subcutaneous weekly injection)

SUMMARY:
The purpose of this multicenter, randomized, placebo-controlled and double-blind study is to evaluate the efficacy and safety of subcutaneous anifrolumab compared with placebo on the overall disease activity in participants with moderate to severe Idiopathic Inflammatory Myopathies (IIM) [polymyositis (PM) or dermatomyositis (DM)] while receiving standard of care (SoC) treatment.

ELIGIBILITY:
Capable of giving informed consent.

Inclusion Criteria:

1. 18 - 75 years old
2. Body weight 40 kg - ≤ 100 kg
3. Must have "probable" or "definite" diagnosis of PM or DM according to the 2017 ACR/EULAR classification criteria for adult myositis.
4. Moderate or severe disease activity per core set measurements.
5. Currently receiving oral prednisone or other polymyositis or dermatomyositis treatments at a stable dose.
6. No history of active tuberculosis or severe COVID-19.
7. Male and female participants must follow contraception guidelines.

Exclusion Criteria:

1. Participants with documented inclusion body myositis (IBM), immune mediation necrotizing myositis (IMNM), juvenile myositis (if diagnosed within 10 years prior to signing the ICF), drug-induced myositis, cancer associated myositis, amyopathic DM, and non inflammatory myopathies (eg, muscular dystrophies).
2. PM and DM patients at a high risk of malignancy.
3. Participants with rapidly progressive interstitial lung disease.
4. Participants with severe muscle damage or permanent weakness due to non-PM or non-DM conditions (i.e. stroke) as per the investigator's opinion.
5. Any history of severe case of herpes zoster infection
6. History of cancer (except adequately treated basal cell carcinoma or cervical cancer in-situ), immunodeficiency, HIV, HBV, active HCV .
7. Any clinical cytomegalovirus or Epstein-Barr virus infection that has not completely resolved within 12 weeks prior to signing the ICF.
8. Opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years prior to randomization.
9. Recent non-opportunistic infection requiring hospitalization or anti-infective treatment.
10. Recent or concurrent enrollment in another clinical study with an investigational product.
11. Lactating, breastfeeding, or pregnant females or females who intend to become pregnant or begin breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-05-14 (Estimated); Study Completion 2028-08-04 (Estimated)

PRIMARY OUTCOMES:
Total Improvement Score (TIS) ≥ 40 response | 52 week
  Participants who have at least moderate improvement in disease activity TIS ≥ 40 and has not met "confirmed deterioration" criteria at 2 consecutive visits

SECONDARY OUTCOMES:
Manual Muscle Testing 8 (MMT-8) (CSM) | 52 week
  MMT-8 (CSM) change from baseline at Week 52.
Oral corticosteroid dose ≤ 7.5 mg/day | 52 week
  Participants who achieve oral corticosteroid dose ≤ 7.5 mg/day at Week 52.
Moderate improvement in disease activity in participants with polymyositis (PM) | 52 week
  Participants with PM who have at least moderate improvement in disease activity (TIS ≥ 40) at Week 52.
Moderate improvement in disease activity in dermatomyositis (DM) participants. | 52 week
  Participants with DM who have at least moderate improvement in disease activity (TIS ≥ 40).
Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) | 8 week
  CDASI activity change from baseline at Week 8 in DM participants only.
Manual Muscle Testing 8 (MMT-8) in PM participants | 52 Week
  MMT-8 change from baseline at Week 52 in PM participants only.
Manual Muscle Testing 8 (MMT-8) in DM participants | 52 Week
  MMT-8 change from baseline at Week 52 in DM participants only.
Core Set Measures (CSMs) | 52 week
  Change from baseline at Week 52 in CSMs:
  * PGA
  * PtGA
  * Muscle enzymes
  * MDAAT extra-muscular disease activity
  * HAQ-DI
Oral corticosteroid dose ≤ 7.5 mg/day in PM participants | 52 week
  PM participants who achieve oral corticosteroid dose ≤ 7.5 mg/day at Week 52
Oral corticosteroid dose ≤ 7.5 mg/day in DM participants | 52 week
  DM participants who achieve oral corticosteroid dose ≤ 7.5 mg/day at Week 52.
Cutaneous Dermatomyositis Activity Investigator Global Assessment (CDA-IGA) | 8, 24, & 52 week
  DM Participants with CDA-IGA ≥ 2 at baseline who achieve:
  * CDA-IGA score ≤ 1 at Week 8 (yes/no)
  * CDA-IGA score ≤ 1 at Week 24 (yes/no)
  * CDA-IGA score ≤ 1 at Week 52 (yes/no)
5-D itch | 8, 24, & 52 week
  DM participants with CDASI activity > 14 at baseline only:
  * 5-D itch change from baseline at Week 8
  * 5-D itch change from baseline at Week 24
  * 5-D itch change from baseline at Week 52
Total Improvement Score (TIS) ≥ 20 Response | 8 week
  Participants who have at least minimal improvement in disease activity TIS ≥ 20 at Week 8 and has not met "confirmed deterioration" criteria at 2 consecutive visits up and including Week 8
Total Improvement Score ≥ 60 Response | 52 week
  Participants who have major improvement in disease activity TIS ≥ 60 at week 52 and has not met "confirmed deterioration" criteria at 2 consecutive visits up to and including Week 52
Cumulative Corticosteroid Use | 24, 52 week
  * Cumulative corticosteroids use as determined by the normalized standardized AUC from baseline up to and including Week 24
  * Cumulative corticosteroids use as determined by the normalized standardized AUC from baseline up to and including Week 52

CONTACTS AND LOCATIONS:
Locations (179):
- United States (32):
  - Research Site, Irvine, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Margate, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Plant City, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Willowbrook, Illinois
  - Research Site, Fairway, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Allen, Texas
  - Research Site, Colleyville, Texas
  - Research Site, El Paso, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Milwaukee, Wisconsin
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Quilmes
  - Research Site, San Miguel de Tucumán
- Australia (5):
  - Research Site, Camperdown
  - Research Site, Nedlands
  - Research Site, New Lambton
  - Research Site, Southport
  - Research Site, Woodville South
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Merksem
- Brazil (7):
  - Research Site, Joinville
  - Research Site, Juiz de Fora
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Haskovo
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Montreal, Quebec
- Chile (4):
  - Research Site, Concepción
  - Research Site, Las Condes
  - Research Site, Osorno
  - Research Site, Santiago
- China (12):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Jining
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Wenzhou
  - Research Site, Zhengzhou
- Research Site, Prague, Czechia
- Denmark (3):
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Odense C
- France (10):
  - Research Site, Angers
  - Research Site, Brest
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (7):
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Freiburg im Breisgau
  - Research Site, Herne
  - Research Site, München
  - Research Site, Tübingen
- Hungary (2):
  - Research Site, Debrecen
  - Research Site, Szeged
- India (11):
  - Research Site, Ahmedabad
  - Research Site, Dehradun
  - Research Site, Gurugram
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, New Delhi
  - Research Site, Puducherry
  - Research Site, Secunderabad
- Israel (5):
  - Research Site, Afula
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
- Italy (11):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Siena
- Japan (14):
  - Research Site, Asahikawa-Shi
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Iruma-Gun
  - Research Site, Kawachinagano-shi
  - Research Site, Kawasaki-shi
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Tachikawa-shi
  - Research Site, Yotsukaido-shi
- Mexico (5):
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
- Research Site, Amsterdam, Netherlands
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Puerto Rico (2):
  - Research Site, Caguas
  - Research Site, San Juan
- South Korea (2):
  - Research Site, Daejeon
  - Research Site, Seoul
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Sabadell
  - Research Site, Valladolid
- Sweden (2):
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (3):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Wolverhampton
- Vietnam (6):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City
  - Research Site, Hồ Chí Minh
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Soares RB, Gabr JB, Ash M, Hosler G. Anifrolumab in Refractory Dermatomyositis and Antisynthetase Syndrome. Case Rep Rheumatol. 2025 Apr 21;2025:5560523. doi: 10.1155/crrh/5560523. eCollection 2025. PMID 40297385